CLINICAL TRIAL: NCT03195959
Title: Effect of Normobaric Hypoxia and Hyperoxia on Pulmonary Hemodynamics in Patients With Pulmonary Hypertension
Brief Title: Effect of Normobaric Hypoxia and Hyperoxia in Patients With Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2016-02136
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial hypertension; Chronic thromboembolic pulmonary hypertension; Hypoxia; Hyperoxia
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PH-Patients: Patients with mean pulmonary artery pressure >25mmHg and a pulmonary arterial wedge pressure <15mmHg during right heart catheterisation, which are diagnosed as having pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension.
  Interventions: Other: Hypoxia and Hyperoxia
- Control group: Patients with clinically indicated right heart catheterisation (because of dyspnea or other signs of PH), but had no PH (no elevated mean pulmonary artery pressure (mPAP <20mmHg)).
  Interventions: Other: Hypoxia and Hyperoxia

INTERVENTIONS:
Other: Hypoxia and Hyperoxia — 10 minutes of breathing a gas mixture with FiO2 0.16 via a tight fitting mask. After 10 minutes of breathing ambient air (normoxia), patients were exposed to hyperoxia (FiO2 1.0) for 10 minutes.

SUMMARY:
Pulmonary Hypertension (PH) is a severe disease with a bad prognosis. However, thanks to extensive research in this field, there are more and better treatment options that allow patients to participate in recreational activities at moderate altitude or bring up the question of air-travel.

Still very few is known about the effects hypoxic conditions have on PH patients. The aim of this study is to investigate the effects of hypoxia in comparison to normoxia and hyperoxia on pulmonary hemodynamics in patients with pulmonary hypertension during routine right heart catheterisation. We aim to get insight into the pathophysiology of pulmonary hemodynamics under hypoxic conditions in comparison to normoxia and hyperoxia in patients with pulmonary arterial and chronic thromboembolic pulmonary hypertension compared with control patients, that are scheduled for right heart catheterisation due to dyspnea but have no PH.

ELIGIBILITY:
Inclusion Criteria:

* clinically indicated right heart catheterisation
* diagnosis of pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension or control without pulmonary hypertension

Exclusion Criteria:

* hemodynamically unstable
* partial pressure of Oxygen < 7.3kPa
* no informed consent
* pulmonary hypertension due to left heart disease, chronic lung disease or miscellaneous (Groups II, III and V) according to Galié ERJ 2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that come to our PH referral center for evaluation of PH and undergo a clinically indicated right heart catheterisation.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change of pulmonary vascular resistance during hypoxia in comparison to normoxia and hyperoxia | Day 1

SECONDARY OUTCOMES:
change of mean pulmonary artery pressure under hyperoxia in comparison to normoxia and hyperoxia | Day 1
change of the cardiac output under hyperoxia in comparison to normoxia and hyperoxia | Day 1
change of the partial pressure of carbon dioxide under hyperoxia in comparison to normoxia and hyperoxia | Day 1
change of the partial pressure of oxygen under hyperoxia in comparison to normoxia and hyperoxia | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, Prof. Dr., Principal Investigator — UniversityHospital Zurich
Locations (1):
- UniversityHospital Zurich, Department of Pulmonology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No